CLINICAL TRIAL: NCT05505084
Title: Comparison of Five Distinct Membranes for Preservation of the Alveolar Ridge Following Tooth Extraction: A Prospective, Randomized, Controlled Clinical Study
Brief Title: Alveolar Ridge Preservation Following Tooth Extraction.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: ZimVie (Industry)
Responsible Party: Principal Investigator, Yucheng Chang, Director of Predoctoral Periodontics, University of Pennsylvania
Other Study IDs: 828879
Record Dates: First submitted 2022-06-01; First posted 2022-08-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Tooth Fractures; Tooth Extraction Status Nos; Caries
Keywords: implant; alveolar ridge preservation
MeSH Terms: conditions — Tooth Fractures | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (5):
- Collatape (Zimmer Dental): This material is a resorbable collagen wound dressing. They are made from bovine Achilles tendons and are a source of Type I collagen. The resorbable wound dressings are sterilized after purification with ethylene oxide.
  Interventions: Procedure: Tooth extraction and ridge preservation using different barrier mermbranes
- Cytoplast Barrier Membranes TXT-200 Singles (Osteogenics Biomedical): Cytoplast Barrier membranes are manufactured from high-density Polytetrafluoroethylene (PTFE) which allows them to withstand exposure to the oral environment. The textured surface increases the surface area available for cellular attachment during dental bone grafting procedures thereby aiding in stabilizing the PTFE membrane. It can be removed non-surgically after at least 21 days.
  Interventions: Procedure: Tooth extraction and ridge preservation using different barrier mermbranes
- Ossix Plus (dantum dental): OssixPlus is a resorbable collagen dental membrane used for Guided Bone Regeneration and Guided Tissue Regeneration. It contains a patented GLYMATRIX cross-linking technology that allows it to maintain barrier functionality for 4 to 6 months. The collagen is derived from porcine.
  Interventions: Procedure: Tooth extraction and ridge preservation using different barrier mermbranes
- Renovix-Plus (Salvin): Renovix Plus is a non-cross-linked extracellular matrix containing Type I, II, and III Collagen, Fibronectin, Laminin, and Elastin. It provides architecture and barrier protection for bone regeneration and soft tissue esthetics. This membrane resorbs within six months.
  Interventions: Procedure: Tooth extraction and ridge preservation using different barrier mermbranes
- BioXclude (Snoasis): BioXclude is a minimally manipulated allograft amnion chorion tissue. It is obtained from consenting mothers who donate their placentas after elective caesarian section delivery. The tissue is processed to cleanse and maintain the tissue. Following processing and dehydration, the allografts are packaged and terminally sterilized.
  Interventions: Procedure: Tooth extraction and ridge preservation using different barrier mermbranes

INTERVENTIONS:
Procedure: Tooth extraction and ridge preservation using different barrier mermbranes — The hopeless and unrestorable teeth are planned for extraction and implant placement.

SUMMARY:
Bone resorption after a tooth extraction is a generally accepted knowledge and has been demonstrated by many animal and human studies. Especially during the first three months followed by the tooth extraction, the volume of bone may change significantly without any interference. Thus, doing a ridge preservation procedure following the extraction is a common standard of care method to maintain the socket volume if implant placement is considered as a treatment option in the future. A variety of materials and methods have been used for ridge preservation. However, it's still inconclusive to determine the best material to maintain the ridge dimension, especially for membrane placement that allows for space maintenance to protect the grafting material. Furthermore, there is no evidence to show any treatment rationale is superior to any other ridge preservation method.

In general, the membrane serves the function of the barrier and space protector. The periodontal surgeon use membranes to exclude the epithelium growth and to limit the collapse of the soft tissue into the healing alveolar socket. Regarding resorbable and non-resorbable membrane materials, both serve the function of protecting the graft material from the oral cavity. However, there are also many demonstrating that without membranes the extraction socket healed nicely without any interferences. The question to us is: Do we need the membrane to exclude the epithelium or any kind of surgical dressing material is sufficient enough to preserve the volume of the extracted ridge?

The object of this study is to compare five popular membranes on the market that present different characteristics of the membranes.

DETAILED DESCRIPTION:
The extraction and the grafting procedure involved in this study are standard of care. The investigators will extract the hopeless teeth and prepare the site for implant placement in 4 months.

The following products will be used during the study:

* Collatape (Zimmer Dental)- approved by the FDA (class III)
* Cytoplast (Osteogenics Biomedical)- cleared by the FDA
* OssixPlus (Dantum Dental)- cleared by the FDA
* Renovix-Plus (Salvin)- cleared by the FDA
* BioXclude (SNOASIS)-certificate from the American Association of Tissue Banking
* PuroⓇ, Zimmer Dental)- cleared by the FDA
* RegenerOssⓇ, Zimmer Dental) - cleared by the FDA

During the appointment for the implant placement. A bone core from all subjects in each treatment group will be collected from the augmentation site instead of drilling away. The sample will be evaluated for the following:

* % viable of bone
* % of connective tissue
* % of residual graft material

ELIGIBILITY:
Inclusion Criteria:

* Subjects must between the ages of 18 and 80.
* Subjects must require removal of at least one maxillary premolar
* Subjects should benefit from an implant-supported crown.
* Subjects must have voluntarily signed the informed consent form.
* Subjects must be assessed as ASA I, ASA II by a member of the research team.

Exclusion Criteria:

* Medical conditions requiring the use of steroids.
* History of leukocyte dysfunction or deficiencies, bleeding deficiencies, renal failure, uncontrolled endocrine disorders, acquired immunodeficiency syndrome or hepatitis.
* History of neoplastic disease requiring the use of chemotherapy or irradiation to head and neck.
* Subjects who have diabetes mellitus.
* Subjects who have undergone administration of any investigational drug or device within 30 days of enrollment in the study.
* Alcohol or drug abuse.
* Subjects who are heavy smokers (greater than 10 cigarettes per day or cigar equivalents) or chew tobacco.
* Conditions or circumstances, in the opinion of the research team, which would prevent completion of study participation or interfere with analysis of study results, such as a history of non-compliance or unreliability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects presenting to the University of Pennsylvania School of Dental Medicine who require extraction of a hopeless tooth due to trauma, caries, or endodontic/periodontal reasons, and who are interested in replacing their tooth with a dental implant.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ridge dimension changes before and after the augmentation. | from the date of the extraction 4 months
  The change in alveolar ridge dimensions will be assessed using CBCT technology after extraction and 4 months after extraction.
Histological Evaluation | 4 months post-augmentation
  A bone core from all subjects in each treatment group will be taken from the augmentation site at the time of implant placement (4 months post-augmentation) and will be evaluated for the composition of the specimen.

SECONDARY OUTCOMES:
Implant site conditions | 4 months post-augmentation
  - Implant stability quotients as determined by resonance frequency analysis.
Implant site conditions | 4 months post-augmentation
  change of the periodontal phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Chang, DMD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Result] Ismail NM, Mustapha MS, Megat R. The subcellular localisation and the time course of bismuth in the gastric mucosa of rats after short-term administration of colloidal bismuth subcitrate. Ann Acad Med Singap. 1997 Nov;26(6):754-7. PMID 9522974
- [Result] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Result] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Result] Misawa M, Lindhe J, Araujo MG. The alveolar process following single-tooth extraction: a study of maxillary incisor and premolar sites in man. Clin Oral Implants Res. 2016 Jul;27(7):884-9. doi: 10.1111/clr.12710. Epub 2015 Nov 14. PMID 26566965
- [Result] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Result] Corbella S, Taschieri S, Francetti L, Weinstein R, Del Fabbro M. Histomorphometric Results After Postextraction Socket Healing with Different Biomaterials: A Systematic Review of the Literature and Meta-Analysis. Int J Oral Maxillofac Implants. 2017 September/October;32(5):1001-1017. doi: 10.11607/jomi.5263. Epub 2017 Feb 23. PMID 28231347
- [Result] Jung RE, Ioannidis A, Hammerle CHF, Thoma DS. Alveolar ridge preservation in the esthetic zone. Periodontol 2000. 2018 Jun;77(1):165-175. doi: 10.1111/prd.12209. Epub 2018 Feb 27. PMID 29484712
- [Result] Bassir SH, Alhareky M, Wangsrimongkol B, Jia Y, Karimbux N. Systematic Review and Meta-Analysis of Hard Tissue Outcomes of Alveolar Ridge Preservation. Int J Oral Maxillofac Implants. 2018 Sep/Oct;33(5):979-994. doi: 10.11607/jomi.6399. PMID 30231083
- [Result] Avila-Ortiz G, Gubler M, Romero-Bustillos M, Nicholas CL, Zimmerman MB, Barwacz CA. Efficacy of Alveolar Ridge Preservation: A Randomized Controlled Trial. J Dent Res. 2020 Apr;99(4):402-409. doi: 10.1177/0022034520905660. Epub 2020 Feb 12. PMID 32050833